CLINICAL TRIAL: NCT01149512
Title: Outcomes of the Adjustable Gastric Band in a Publicly Funded Obesity Program
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Daniel Birch, MSc, MD, FRCSC, FACS, University of Alberta
Other Study IDs: Pro00014271
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LAGB patients in Weight Wise Program: All patients seen within the Weight Wise program and selected for surgical management, who have undergone LAGB will be included in this analysis.

SUMMARY:
The majority of data documenting the outcomes for the adjustable gastric band (LAGB) originate from non-publicly funded surgical centres. The investigators aim to investigate the clinical outcomes of LAGB from a publicly funded Canadian obesity management program. This program recognized obesity as a chronic disease, providing extensive pre-operative multidisciplinary assessment and long term patient follow-up. Patients are selected for surgical management carefully by a multidisciplinary team and the LAGB is presented as one option to surgical management. Further, the investigators will investigate the operational impacts, including direct and indirect costs related the LAGB, to determine long term impacts on publicly funded hospitals within Canada.

ELIGIBILITY:
Inclusion Criteria:

* All patients seen within the Weight Wise program and selected for surgical management, who have undergone LAGB will be included in this analysis.

Exclusion criteria:

* Patients who have undergone selection for surgery outside this process, or who have had surgery elsewhere.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients seen within the Weight Wise program and selected for surgical management, who have undergone LAGB will be included in this analysis.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for the Advancement of Minimally Invasive Surgery & Weight Wise Program, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LAGB Patients in Weight Wise Program
Started | 178
Completed | 178
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LAGB Patients in Weight Wise Program
Number analyzed (Participants) | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153
  Male | 25
initial BMI [Mean (Standard Deviation); unit: kg/m^2] | 44.2 (7)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Total Body Weight Loss
Description: the percent total body weight loss between Baseline and 1 year the percent total body weight loss between Baseline and 2 years the percent total body weight loss between Baseline and 3 years
Time Frame: baseline to 1 year, baseline to 2 years, baseline to 3 years
Population: Three patients' weight data were not included in the weight loss analysis owing to early removal of band (n = 1) and complication or pregnancy affecting weight (n = 2) before 1-year follow-up. 79 patients reached 2 year follow up time point and 38 patients reached 3 year follow up time point.
Measure: Mean (Standard Deviation); unit: % of total body weight loss
Arm/Group | LAGB Patients in Weight Wise Program
Number analyzed (Participants) | 175
% of total body weight loss
  Baseline to 1 year | 15.8 (7.6)
  Baseline to 2 years: number analyzed (Participants) | 79
  Baseline to 2 years | 20.7 (11)
  Baseline to 3 years: number analyzed (Participants) | 38
  Baseline to 3 years | 20.3 (10)

2. Secondary Outcome: % of Excess Body Weight Loss
Description: the percent of excess body weight loss between Baseline and 1 year the percent of excess body weight loss between Baseline and 2 years the percent of excess body weight loss between Baseline and 3 years
Time Frame: baseline to 1 year, baseline to 2 years, baseline to 3 years
Population: 3 not included the same reason as above.
Measure: Mean (Standard Deviation); unit: % of excessive weight loss
Arm/Group | LAGB Patients in Weight Wise Program
Number analyzed (Participants) | 175
% of excessive weight loss
  Baseline to 1 year | 34.1 (16)
  Baseline to 2 years: number analyzed (Participants) | 79
  Baseline to 2 years | 44 (23)
  Baseline to 3 years: number analyzed (Participants) | 38
  Baseline to 3 years | 43.4 (21)

ADVERSE EVENTS:
Time Frame: 3-year follow-up
Arm/Group | LAGB Patients in Weight Wise Program
Serious Adverse Events (participants affected / at risk) | 0/178
Other Adverse Events (participants affected / at risk) | 50/178
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAGB Patients in Weight Wise Program (N=178)
postoperative nausea (Gastrointestinal disorders) | 34 (34)
band migration (Surgical and medical procedures) | 10 (10)
port site complications (Surgical and medical procedures) | 2 (2)
band leakage (Surgical and medical procedures) | 2 (2)
incisional hernia (Surgical and medical procedures) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No